CLINICAL TRIAL: NCT00331227
Title: Effect of Supplemental Flavonoids on Endothelial Function, Lipids, and Markers of Inflammation
Brief Title: Flavonoid Supplementation and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 202021
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2007-03

CONDITIONS: Healthy
Keywords: flavonoids; food supplements; endothelial function; no conditions allowed, healthy volunteers only

INTERVENTIONS:
Drug: Isotonix OPC-3 (flavonoid supplement)

SUMMARY:
Flavonoids are one of the many classes of natural chemicals found in a variety of foods. People with the highest flavonoid blood levels have the lowest rates of coronary heart disease. This is considered one of the reasons why high fruit and vegetable consumption is associated with lower rates of heart disease, although it is not known if taking a flavonoid supplement provides the same protection as eating fruits and vegetables.

The purpose of this study is to determine if a particular flavonoid supplement, called Isotonix OPC-3, taken on a daily basis, will improve the function of arterial vessels. Arteries normally constrict after eating a high-fat meal. This study will examine the potential of the OPC-3 to lessen this constriction response. Approximately 25 people will be involved in this research project and participation will last for 10 weeks.

DETAILED DESCRIPTION:
We propose to use a supplement made by NutraMetrix (called OPC-3), consisting of oligomeric proanthocyanidins derived from grape seed, pine bark, bilberry, citrus and red wine extracts, to determine effects on endothelial function, lipoproteins and inflammation. The primary outcome measure will be endothelial function as assessed by digital response to hyperemia using peripheral arterial tonometry, measured both in the fasting state and after a single standardized high-fat meal, when transient dysfunction is expected to occur. Secondary outcome measures will be the lipid profile, hs-CRP, and Lp-PLA2. The recruitment population will be healthy volunteers. The design will be a randomized, placebo-controlled, double-blind, cross-over trial lasting 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age or older
* no pregnant potential

Exclusion Criteria:

* History of coronary artery disease
* History of cerebrovascular disease
* History of heart failure
* Diabetes
* Renal impairment
* Uncontrolled hypertension
* Untreated or clinically evident thyroid disease
* Currently taking medications or supplements with known or potential lipid-altering effects including: phytosterols, statins, cholestin, niacin, fibrates, psyllium fiber, bile acid sequestrants, diabetic medications, and weight control medications such as orlistat
* Pregnancy or breastfeeding
* Tobacco use - Participants will be excluded with a history of smoking anytime in the past 6 months.
* Inappropriate for participation in a study, if in the opinion of the investigator it is questionable whether the participant will be able to comply with all aspects of the protocol (e.g. inadequate cognitive skills, possible drug abuse or dependence, suspected psychiatric problems, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-05; Study Completion 2006-12

PRIMARY OUTCOMES:
Change in endothelial function from baseline

SECONDARY OUTCOMES:
CRP
Lipid profile
Lp-PLA2

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Barringer, MD, Principal Investigator — Carolinas Medical Center